CLINICAL TRIAL: NCT05124015
Title: Exercise Capacity Respiratory Muscle Strength Pulmonary Function Dyspnea and Physical Activity in Pediatric Pulmonary Arterial Hypertension
Brief Title: Exercise Capacity Respiratory Muscle Strength Dyspnea and Physical Activity in Pediatric Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi University 128
Record Dates: First submitted 2021-11-15; First posted 2021-11-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: muscle strength; exercise; exercise test; physical activity; pulmonary arterial hypertension; Respiratory Function Tests
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with pulmonary arterial hypertension: Exercise capacity using six minute walk test, respiratory muscle strength using mouth pressure device, pulmonary function using spirometry, dyspnea using Modified Borg scale physical activity using multi-sensor activity monitor.
- Healthy controls: Exercise capacity using six minute walk test, respiratory muscle strength using mouth pressure device, pulmonary function using spirometry, dyspnea using Modified Borg scale physical activity using multi-sensor activity monitor.

SUMMARY:
The primary aim of this study was to evaluate exercise capacity, respiratory muscle strength, pulmonary function, dyspnea and physical activity levels in pediatric PAH patients and compare them with healthy controls.

The secondary aim of the study was; To investigate the relationship of dyspnea with exercise capacity, respiratory muscle strength, respiratory functions, physical activity and blood count parameters in pediatric PAH patients.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a mean pulmonary artery pressure of 25 mmHg or more at rest. Since the diagnosis of PAH can be made mostly in the late phase of the disease, severe functional and hemodynamic problems are prevalent in patients. In addition, patients commonly present with dyspnea, fatigue, weakness, general exercise intolerance, chest pain, syncope, and abdominal distension. These signs and symptoms are due to reduced oxygen consumption and decreased cardiac output. Activity dyspnea is evident in patients in the early stages of the disease. There is limited number of studies in pediatric PAH patients investigating exercise intolerance. While the cardiopulmonary exercise test can be safely performed in pediatric PAH patients, the six-minute walk test is both an independent predictor of prognosis and reflects the severity of the disease in these patients. However, there are no studies in the literature investigating and comparing exercise capacity, respiratory muscle strength, respiratory functions, dyspnea, and physical activity levels in pediatric PAH patients compared to age- and sex-matched healthy children. For this reason, in this study, the level of physical impairments of children with pediatric PAH was investigated for the first time compared to healthy children. In addition, there has been no study in the literature investigated the relationship between dyspnea, which can be seen significantly from the early stages of the disease in pediatric PAH patients, with exercise capacity, respiratory function, respiratory muscle strength, physical activity levels and blood count parameters.

It is a cross-sectional study. At least 15 PAH patients and 15 age-and sex-matched healthy controls were aimed to include in the study. Individuals' exercise capacity using six minute walk test, respiratory muscle strength using a mouth pressure device, pulmonary function using spirometry, dyspnea using Modified Borg scale, physical activity using multi-sensory activity monitor were evaluated. The assessments were completed in two days.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for patients with PAH are as follows:

1. Between the ages of 6-18
2. Diagnosed with pulmonary arterial hypertension
3. Clinically stable and receiving standard medical treatment

The inclusion criteria for healthy children are as follows:

1) To be between the ages of 6-18

Exclusion Criteria:

The exclusion criteria for patients with PAH are as follows:

1) Having any acute infection, orthopedic, neurological, cooperation, vision or hearing problems that may interfere during the measurements

The exclusion criteria for healthy children are as follows:

1. Having any acute or chronic illness
2. Active or ex-smoker

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 13 patients with PAH and 15 healthy individuals were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | First Day
  Functional exercise capacity was evaluated using the 6- Minute Walk Test. 6- Minute Walk Test will be applied according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.

SECONDARY OUTCOMES:
Respiratory muscle strength | First Day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were measured using a portable mouth pressure measuring device according to ATS and ERS criteria.
Pulmonary function (Forced vital capacity (FVC)) | First Day
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, forced vital capacity (FVC)was evaluated.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First day
  Pulmonary function was evaluated with the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, forced expiratory volume in the first second (FEV1) was evaluated.
Pulmonary function (FEV1 / FVC) | First day
  Pulmonary function was evaluated with the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, FEV1 / FVC was evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%)was evaluated.
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, peak flow rate (PEF) was evaluated.
Dyspnea | First day
  Subjectively, dyspnea at rest and during activity, orthopnea, paroxysmal nocturnal dyspnea, activities that increase dyspnea, and severity of dyspnea (using the Modified Borg scale) was evaluated.
Physical activity (Total energy expenditure) | Second Day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day)) | Second Day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity time (min / day)) | Second day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent (MET / day)) | Second day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps (steps / day)) | Second day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Time spent lying down (min / day) days)) | Second day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep time (min / day)) | Second day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Baytok, Pt. MSc, Study Chair — Gazi University, Faculty of Health Sciences, Department of Cardiopulmonary Physical Therapy and Rehabilitation; Gülşah Barğı, PhD. Pt., Principal Investigator — Izmir Democracy University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Betül Yoleri, Pt. MSc, Principal Investigator — Gazi University, Faculty of Health Sciences, Department of Cardiopulmonary Physical Therapy and Rehabilitation; Fatma İncedere, Dr, Principal Investigator — Gazi University; Serdar Kula, Prof.Dr., Principal Investigator — Gazi University; Fatma Sedef Tunaoğlu, Prof.Dr., Principal Investigator — Gazi University; Meral Boşnak Güçlü, Prof. Dr., Study Director — Gazi University, Faculty of Health Sciences, Department of Cardiopulmonary Physical Therapy and Rehabilitation
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Background] McGoon M, Gutterman D, Steen V, Barst R, McCrory DC, Fortin TA, Loyd JE; American College of Chest Physicians. Screening, early detection, and diagnosis of pulmonary arterial hypertension: ACCP evidence-based clinical practice guidelines. Chest. 2004 Jul;126(1 Suppl):14S-34S. doi: 10.1378/chest.126.1_suppl.14S. PMID 15249493
- [Background] Douwes JM, Hegeman AK, van der Krieke MB, Roofthooft MT, Hillege HL, Berger RM. Six-minute walking distance and decrease in oxygen saturation during the six-minute walk test in pediatric pulmonary arterial hypertension. Int J Cardiol. 2016 Jan 1;202:34-9. doi: 10.1016/j.ijcard.2015.08.155. Epub 2015 Aug 28. PMID 26386916
- [Background] Cappelleri JC, Hwang LJ, Mardekian J, Mychaskiw MA. Assessment of measurement properties of peak VO(2) in children with pulmonary arterial hypertension. BMC Pulm Med. 2012 Sep 10;12:54. doi: 10.1186/1471-2466-12-54. PMID 22963001
- [Background] Smith G, Reyes JT, Russell JL, Humpl T. Safety of maximal cardiopulmonary exercise testing in pediatric patients with pulmonary hypertension. Chest. 2009 May;135(5):1209-1214. doi: 10.1378/chest.08-1658. Epub 2008 Dec 31. PMID 19118264